CLINICAL TRIAL: NCT02183389
Title: Relative Bioavailability of a Single Oral Dose of Warfarin (10 mg qd) After Coadministration With Multiple Oral Doses of BI 1356 (5 mg qd) Compared to the Bioavailability of a Single Oral Dose of Warfarin (10 mg qd) Alone in Healthy Male Volunteers (an Open Label, Two Periods, Fixed-sequence, Clinical Phase I Study)
Brief Title: Bioavailability of Warfarin After Coadministration With Multiple Doses of BI 1356 Compared to the Bioavailability of Warfarin Alone in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1218.28
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Warfarin; Linagliptin

ARMS (2):
- Treatment B: BI 1356 and Warfarin (Experimental): BI 1356 for 12 days combined with a single dose of warfarin on day 6
  Interventions: Drug: Warfarin; Drug: BI 1356
- Treatment A: Warfarin (Active Comparator): Warfarin as single dose
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Warfarin
Drug: BI 1356
  Arms: Treatment B: BI 1356 and Warfarin

SUMMARY:
To investigate whether and to what extent BI 1356 affects pharmacokinetic and pharmacodynamic parameters of warfarin

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria:

  * Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
* Age ≥ 18 and Age ≤ 50 years
* BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and the local legislation
* Homozygote wild-type carriers (*1/*1) of cytochrome P 450 (CYP) 2C9

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for Torsades de points (TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Exclusion criteria specific for this study:

* Anemia at screening
* Galactose intolerance
* Lactase deficiency
* Glucose-galactose-malabsorption

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 168 hours after start of study medication
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 168 hours after start of study medication

SECONDARY OUTCOMES:
Area under the concentration time curve (AUC) of the analyte in plasma at different time points | Up to 168 hours after start of study medication
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | Up to 168 hours after start of study medication
Terminal rate constant in plasma (λz) | Up to 168 hours after start of study medication
Terminal half life of the analyte in plasma (t1/2) | Up to 168 hours after start of study medication
Mean residence time of the analyte in the body after p.o. administration (MRTpo) | Up to 168 hours after start of study medication
Apparent clearance of the analyte in the plasma after extravascular administration (CL/F) | Up to 168 hours after start of study medication
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F) | Up to 168 hours after start of study medication
Number of patients with adverse events | Up 42 days
Number of patients with relevant changes in physical examination | Up to 14 days after last study drug administration
Number of patients with relevant changes in vital signs (Blood Pressure (BP), Pulse Rate (PR)) | Up to 14 days after last study drug administration
Number of patients with relevant changes in 12-lead resting electrocardiogram (ECG) | Up to 14 days after last study drug administration
Number of patients with relevant changes in laboratory values | Up to 14 days after last study drug administration
Assessment of tolerability a 4-point scale by the investigator | Up 42 days
International normalised ratio, area under the concentration time curve of the analyte in plasma over the time interval from time zero to 168 hours (INR AUC0-168) | Up to 168 hours after start of treatment
International normalised ratio, maximum concentration of the analyte in plasma (INRmax) | Up to 168 hours after start of treatment
Prothrombin time, area under the concentration time curve of the analyte in plasma over the time interval from time zero to 168 hours (PT AUC0-168) | Up to 168 hours after start of treatment
Prothrombin time, maximum concentration of the analyte in plasma (PTmax) | Up to 168 hours after start of treatment